CLINICAL TRIAL: NCT05275725
Title: Finding Solutions to Thrive After Birth Asphyxia in Africa: An Open-label Dose-finding Clinical Trial (Phase Ib Study)
Brief Title: Finding Solutions to Thrive After Birth Asphyxia in Africa
Acronym: SANE-Uganda
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pia Wintermark (Other)
Collaborators: Kawempe National Referral Hospital (Unknown); Saint Francis Hospital (Other); Walimu (Other)
Responsible Party: Sponsor-Investigator, Pia Wintermark, Associate Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SANE-Uganda
Record Dates: First submitted 2022-02-08; First posted 2022-03-11 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Birth Asphyxia
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Phase Ib open-label single-arm dose-finding clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sildenafil (Experimental)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Dose group 1st dose 2nd dose 3rd dose 4-14th doses Treatment Total dose/day frequency dose/day Group 1: #1-14=2 mg/kg q12h (4 mg/kg/day) Group 2: #1 = 2 mg/kg, #2-14 = 2.5 mg/kg q12h (5 mg/kg/day) Group 3: #1 = 2 mg/kg, #2 = 2.5 mg/kg, #3-14 = 3 mg/kg q12h (6 mg/kg/day) Group 4: #1 = 2.5 mg/kg, #2-14 = 3 mg/kg q12h (6 mg/kg/day) Group 5: #1-14 = 3 mg/kg q12h (6 mg/kg/day)

SUMMARY:
Neonatal encephalopathy (NE) is the third leading cause of under 5-year mortality and contributes substantially to long-term neurological morbidity worldwide. In low-income countries (LICs), families often lack the resources to care for affected children. For those with disabilities, stigma is high, and social and emotional impacts are substantial. Improving our understanding of NE in LICs is crucial if intervention strategies are developed. Providing access to an affordable and easy-to-administer treatment after birth may improve survival, early brain development and later outcome, maximizing developmental potential.

The primary objective of this study is to investigate the feasibility, safety and tolerability of administering sildenafil as a neuroprotective/neurorestorative strategy to improve early brain development in a cohort of children with NE in Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Male and female neonates meeting the criteria for birth asphyxia
* Gestational age ≥ 36 weeks and birth weight ≥ 1800 g;
* Admitted to Kawempe Hospital or Nsambya Hospital within 48 hours of life;
* Need for continued resuscitation after birth and/or 5-minute Apgar score ≤5;
* Evidence of neonatal encephalopathy by an abnormal neurological exam (modified Sarnat score of 2-3 or abnormal aEEG).

Exclusion Criteria:

* Absent heart rate at 10 minutes/imminent death
* Neonates with major congenital malformations
* Neonates with grade 3 AKI (serum creatinine rise ≥3x lowest previous creatinine or creatinine > 2.5 mg/dL = 221 mcmol/L or receipt of dialysis)
* Neonates with intraventricular and/or intraparenchymal hemorrhage on cranial ultrasound (cUS) performed on day 1-2 of life
* Mother living permanently outside 20km radius of Kawempe Hospital or Nsambya Hospital
* Neonates whose parents are unwilling or unable to give informed written consent to enter the study

Ages: 0 Days to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerable dose of sildenafil | within 30 days of drug administration

SECONDARY OUTCOMES:
Incidence of adverse events (Safety and Tolerability) | within 30 days of drug administration
  safety, assessed through the reporting of adverse events, such as death, hypotension, persistent pulmonary hypertension, altered hepatic function, seizures, intraventricular and/or intraparenchymal hemorrhage
Sildenafil concentrations | within 30 days of drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Kawempe National Referral Hospital, Kawempe, Uganda

IPD SHARING:
Plan to Share IPD: No
No individual participant data sharing